CLINICAL TRIAL: NCT01968798
Title: ASPREE Cancer Endpoints Study
Acronym: ACES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Aging (NIA) (NIH); Monash University (Other); Berman Center for Outcomes and Clinical Research (Other); National Health and Medical Research Council, Australia (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3U01AG029824-02S1 (NIH)
Record Dates: First submitted 2013-09-19; First posted 2013-10-24 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Cancer
Keywords: ACES; ASPREE Cancer Endpoints Study; Cancer; Aspirin; Tumor
MeSH Terms: conditions — Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): 100 mg enteric-coated aspirin
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 100mg enteric-coated aspirin, taken daily
  Arms: Aspirin
Drug: Placebo — 100mg enteric-coated placebo, taken daily
  Arms: Placebo

SUMMARY:
The ASPREE Cancer Endpoint Study (ACES), an ancillary study of the ASPirin in the Prevention of Events in the Elderly (ASPREE) Study, will allow for the examination of the effect of daily low-dose aspirin (100 mg) compared to placebo, on specific DNA biomarkers and selected specific incident and recurrent cancer and metastases. The establishment of this ACES biobank will allow for the exploration of DNA-related molecular mechanisms of aspirin's protective effect against cancer, cancer associated mortality and metastases, using blood or saliva DNA specimens, urine, and tumor tissue.

DETAILED DESCRIPTION:
The ASPREE Cancer Endpoint Study (ACES) is an ancillary study of the ASPirin in the Prevention of Events in the Elderly (ASPREE) Study, a 5 year randomized placebo- controlled trial of 100 mg of daily aspirin in 19,000 elderly in Australia and the US to determine whether the benefits of low dose daily aspirin outweigh the bleeding risks. The primary outcome of ASPREE is defined as prolongation of "disability-free life", measured as survival without physical disability or dementia. At present, the primary purpose of ACES is to: 1) collect information about participant cancer screenings, cancer diagnosis, and family history of cancer and to 2) establish a biologic specimen repository (biobank) for DNA and tumor tissue, and urine from the ASPREE large healthy aging population in the US and Australia for future use by ASPREE, NIA and NCI investigators, and academicians from the broader research community. At a time in the future and under separate application, the stored blood or saliva, urine, and tumor tissue, together with other information obtained about these participants (in relation to their health, lifestyle and other circumstances) will be analyzed to address specific questions regarding the association of biomarkers and major health outcomes including cancer.

ELIGIBILITY:
Open Only to Participants in Parent ASPREE study

1. Inclusion criteria: Men and women 65 years and older in US (African American or Hispanic), and 70 years of age and over in Australia (Caucasian, Asian, other minorities). Based on NIAs discretion, select US sites may be recruiting Caucasians 70 and older or 75 and older.
2. Exclusion criteria: (please see www.ASPREE.org for more detailed list of exclusion criteria) i. History of diagnosed dementia or score < 78 on the Modified Mini Mental State Exam at the second pre-randomization (baseline) visit.

   ii. Disability, defined as dependence in one or more Katz activity of daily living.

   iii. Cardiovascular events, intercurrent illness likely to cause death within the next 5 years, a current or recurrent condition with a high risk of major bleeding, e.g. cerebral aneurysm, cerebral AV malformation, any bleeding diathesis, recent peptic ulcer and liver disease.

   iv. Anemia, i.e. hemoglobin level below the normal value (males: 12 g/dL, females: 11 g/dL).
3. Participants eligible for the ASPREE Cancer Endpoints Study (ACES) include any participants recruited into the parent ASPREE study in the United States and Australia. ACES participants will be asked to consent to:

i. Collection and storage of blood or saliva DNA samples and urine and data for future use. If ASPREE participants are unwilling to contribute biological samples, this will not in any way jeopardize their continued enrolment in ASPREE.

ii. Collection of cancer tumor specimens and storage and data for future use.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14500 (Estimated)
Dates: Start 2013-09; Primary Completion 2019-01 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of daily low-dose aspirin (100 mg) compared to placebo, on specific DNA biomarkers and selected specific incident and recurrent cancer and metastases. | every 6 months
  The ASPREE Cancer Endpoint Study (ACES) will allow for the examination of the effect of daily low-dose aspirin (100 mg) compared to placebo, on specific DNA biomarkers and selected specific incident and recurrent cancer and metastases. The establishment of this ACES biobank will allow for the exploration of DNA-related molecular mechanisms of aspirin's protective effect against cancer, cancer associated mortality and metastases, using blood or saliva DNA specimens, urine, and tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Murray, MD, MSc, Principal Investigator — Berman Center
Locations (40):
- United States (40):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Howard University, Washington D.C., District of Columbia
  - University of Florida Department of Aging and Geriatrics, Gainesville, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory/ Atlanta VAMC, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Baton Rouge General, Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Our Lady of the Lake Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins St. Tammany Parish Hospital, Covington, Louisiana
  - Mary Bird Perkins Terrebonne General Hospital, Houma, Louisiana
  - LSU Health Sciences- New Orleans, New Orleans, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - LSU Health Sciences- Shreveport, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Detroit Clinical Research Center, Novi, Michigan
  - HealthPartners Research Institute, Minneapolis, Minnesota
  - Phalen Village Clinic, Saint Paul, Minnesota
  - Central Jersey Medical Center, Elizabeth, New Jersey
  - New Jersey Medical College, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - Queens Cancer Medical Center, Queens, New York
  - Wake Forest University Baptist Medical Center, Greensboro, North Carolina
  - The Brody School of Medicine at ECU, Greenville, North Carolina
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Health Sciences Research Center, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of TX Medical Branch, Galveston, Texas
  - Regional Academic Health Center, Harlingen, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: Public ASPREE website — http://www.aspree.org